CLINICAL TRIAL: NCT03579199
Title: Practical Application of Indocyanine Green Camera in Laparoscopic Liver Surgery
Acronym: CAMVIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: FLUOPTICS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P170105J; 2017-A02807-46 (Other: N° IDRCB)
Record Dates: First submitted 2018-05-25; First posted 2018-07-06 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Liver Tumor
Keywords: hepatic tumor; liver; ICG; ICG camera; laparoscopy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exploration of abdominal cavity using a NIR/ICG camera (Experimental)
  Interventions: Device: exploration of abdominal cavity and liver using a NIR/ICG camera

INTERVENTIONS:
Device: exploration of abdominal cavity and liver using a NIR/ICG camera — exploration of abdominal cavity and liver using a NIR/ICG camera

SUMMARY:
"Indocyanine Green (ICG) is a dye used as an indicator of hepatic function considering its capacity to be eliminated only by the bile. Thus, ICG tend to remain in liver tumors.

The hypothesis of CAMVIC study is that the use of fluorescence imaging during laparoscopic hepatic surgery will allow to detect small subcapsular superficial lesions undetected by other diagnostic methods, which will improve the results of the oncologic treatment."

DETAILED DESCRIPTION:
"Thanks to the property of ICG to release a fluorescent signal when excited by a Near Infra Red (NIR) light source, ICG fluorescence has been widely used during several clinical situations (angiography, lymphography,..). Few years ago it has been shown that hepatic tumors could be seen with a NIR camera able to view ICG fluorescence thanks to the depot in or around the tumor of the dye injected during preop.Since, this fluorescence imaging technique potential has been underlined to identify tumors undiagnosed before surgery. Pre-operative examination of hepatic lesions is based on 3 points:

* visual examination
* two-hand palpation
* intra-operative ultrasound.

During laparoscopic hepatic surgery it is not possible to palpate the liver thus peroperative examination of the liver surface is harder than during open surgery. Moreover per-operative ultrasound is not a reliable tool in order to explore liver surface. However the latest development of NIR cameras able to view ICG fluorescence could add a benefit in laparoscopic surgery in view of its capacity to detect superficial lesions, even those of small dimension."

ELIGIBILITY:
Inclusion Criteria:

* men and woman aged of 18 yo and more
* patients with liver tumor
* patient affiliated to french social security

Exclusion Criteria:

* Patient unable to give a signed informed consent
* patient under guardianship or curator
* patient deprived of liberty by judicial or administrative decision or placed under judicial protection
* patient refusing to undergo the specific technique
* pregnant or lactating women
* patient with icteric cholestasis
* patient with contraindication to coelioscopy
* patient with known allergy to cyanines
* patient who must undergo staged hepatectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
number of superficial nodules detected with the device during peroperative examination compared to the number of superficial nodules detected during preoperative imaging and new surface nodules detected at 6 month postoperative imaging | through study completion, an average of 6 months
  sensitivity will be assessed by the number of superficial nodules detected with the device during peroperative examination compared to the number of superficial nodules detected during preoperative imaging and new surface nodules detected at 6 month postoperative imaging
Histological analysis of explanted liver parts | 1 month
  histological analysis will indicate the nature of the explanted part: tumoral tissue or healthy tissues. Results will be obtained during the month following the hepatectomy

SECONDARY OUTCOMES:
bilirubin and prothrombin levels | at Day 1, day 3 and day 5 visits
  predictive value of the fluorescence dynamic on postoperative hepatic function will be assessed with bilirubin and prothrombin levels at day 1, day 3 and day 5 visits

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hépato Biliaire de l'hopital Paul Brousse, Villejuif, France

IPD SHARING:
Plan to Share IPD: No